CLINICAL TRIAL: NCT04414163
Title: An Open-label, Single-arm, Phase 2 Study to Investigate the Efficacy and Safety of IMC-001 in Patients With Relapsed or Refractory Extranodal NK/T Cell Lymphoma, Nasal Type
Brief Title: A Study of IMC-001 in Subjects With Relapsed or Refractory Extranodal NK/T Cell Lymphoma, Nasal Type
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneOncia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMC-001-201
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type; Extranodal NK/T-cell Lymphoma
Keywords: IMC-001; IMC-001-201; DISTINKT
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — IMC-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMC-001 (Experimental): Single Dose level (IMC-001 20mg/kg, every 2 weeks)
  Interventions: Drug: IMC-001

INTERVENTIONS:
Drug: IMC-001 — Single dose level for enrollment subject (IMC-001 20mg/kg every 2 weeks)
  Other Names: Not confirm yet

SUMMARY:
This is a phase 2, Open-label, to investigate the efficacy and safety of IMC-001 in patients with Relapsed or Refractory extranodal NK/T cell lymphoma, nasal type

DETAILED DESCRIPTION:
IMC-001 is a PD-L1 targeting, fully human monoclonal antibody. The purpose of this study is to determine and evaluate the efficacy and safety of IMC-001. 20mg/kg every 2 weeks, IV infusion of IMC-001 will be tested in subjects with Relapsed or Refractory extranodal NK/T cell lymphoma, nasal type.

ELIGIBILITY:
Inclusion Criteria:

1. ENKTL diagnosis;

   * Histologically confirmed diagnosed with extranodal NK/T-cell lymphoma, nasal type
   * At least 1 previous line of systemic therapy
   * Documented disease progression of last therapy
2. Adult age(as defined by respective country)
3. The nature of the study and voluntarily sign an ICF
4. ECOG 0 or1
5. Adequate hematologic function, hepatic function, and renal function

Exclusion Criteria:

1. Previously treated with an anti-PD-L1 or anti-PD-1 antibody
2. Known presence of symptomatic CNS metastases
3. Prior allogeneic HSCT or solid organ transplantation
4. Any active autoimmune disease or a documented history of autoimmune disease
5. Apparent active or latent TB and known viral infection with hepatitis B virus or hepatitis C virus
6. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Objective Response Rate(ORR) | through study completion, an average of 1 year
  Lugano criteria with LYRIC modification

SECONDARY OUTCOMES:
Evaluate safety of IMC-001 | through study completion, an average of 1 year
  Terms, frequency, severity and seriousness of AEs and relationship of AEs to IMC-001
Evaluate additional efficacy variables of IMC-001 : Complete Response (CR) rate | The imaging assessment will be performed every 12 weeks (± 1 week) according to the Lugano criteria with LYRIC modification by centralized independent review, and the Lugano criteria with LYRIC modification and the Lugano Criteria by investigator.
  Complete Response (CR) rate, (Unit of Measure: Percentage of participants)
  1. Variables determined by the centralized independent assessment per the Lugano criteria with LYRIC modification
  2. Variables determined by the investigator assessment per the Lugano criteria with LYRIC modification
  3. based on response as determined by the investigator per the Lugano criteria
Evaluate additional efficacy variables of IMC-001 : Disease Control Rate (DCR) | The imaging assessment will be performed every 12 weeks (± 1 week) according to the Lugano criteria with LYRIC modification by centralized independent review, and the Lugano criteria with LYRIC modification and the Lugano Criteria by investigator.
  Disease Control Rate (DCR), (Unit of Measure: Percentage of participants)
  1. Variables determined by the centralized independent assessment per the Lugano criteria with LYRIC modification
  2. based on response as determined by the investigator per the Lugano criteria
Evaluate additional efficacy variables of IMC-001 : Progression-Free Survival (PFS) | The imaging assessment will be performed every 12 weeks (± 1 week) according to the Lugano criteria with LYRIC modification by centralized independent review, and the Lugano criteria with LYRIC modification and the Lugano Criteria by investigator.
  Progression-Free Survival (PFS), (Unit of Measure: Months)
  1. Variables determined by the centralized independent assessment per the Lugano criteria with LYRIC modification
  2. Variables determined by the investigator assessment per the Lugano criteria with LYRIC modification
  3. based on response as determined by the investigator per the Lugano criteria
Evaluate additional efficacy variables of IMC-001 : Duration of Response (DOR) | The imaging assessment will be performed every 12 weeks (± 1 week) according to the Lugano criteria with LYRIC modification by centralized independent review, and the Lugano criteria with LYRIC modification and the Lugano Criteria by investigator.
  Duration of Response (DOR), (Unit of Measure: Months)
  1. Variables determined by the centralized independent assessment per the Lugano criteria with LYRIC modification
  2. based on response as determined by the investigator per the Lugano criteria
Evaluate additional efficacy variables of IMC-001 : Time to Progression (TTP) | The imaging assessment will be performed every 12 weeks (± 1 week) according to the Lugano criteria with LYRIC modification by centralized independent review, and the Lugano criteria with LYRIC modification and the Lugano Criteria by investigator.
  Time to Progression (TTP), (Unit of Measure: Months)
  1. Variables determined by the centralized independent assessment per the Lugano criteria with LYRIC modification
  2. based on response as determined by the investigator per the Lugano criteria
Evaluate additional efficacy variables of IMC-001 : Overall Response Rate (ORR) | The imaging assessment will be performed every 12 weeks (± 1 week) according to the Lugano criteria with LYRIC modification by centralized independent review, and the Lugano criteria with LYRIC modification and the Lugano Criteria by investigator.
  Overall Response Rate (ORR), (Unit of Measure: Percentage of participants)
  1. Variables determined by the investigator assessment per the Lugano criteria with LYRIC modification
  2. based on response as determined by the investigator per the Lugano criteria
Evaluate additional efficacy variables of IMC-001 : Overall Survival (OS) | through study completion, an average of 1 year
  Overall Survival (OS), (Unit of Measure: Months)
Determine the pharmacokinetic (PK) profile of IMC-001 : Ctrough | Cycle 1 Day 1(Pre-dose/EOI + 1 hr ± 5 min), Cycle 2, 4, 7, 10, 13 Day 1(Pre-dose up to 1 hr before/EOI + 1 hr ± 5 min) (each cycle is 14 days)
  The trough level or trough concentration (Ctrough) of IMC-001 measured at specified time points.
Determine the pharmacokinetic (PK) profile of IMC-001 : Cmax | Cycle 1 Day 1(Pre-dose/EOI + 1 hr ± 5 min), Cycle 2, 4, 7, 10, 13 Day 1(Pre-dose up to 1 hr before/EOI + 1 hr ± 5 min) (each cycle is 14 days)
  The maximum observed serum concentration (Cmax) of IMC-001 observed during dosing interval.
Characterize the immunogenicity of IMC-001 : Incidence of Anti-Drug Antibodies (ADA) | Screening, prior to infusion at Cycle 4, 7, 10, and 13, End of Treatment, Safety Follow up (each cycle is 14 days, EOT: 28-day (+ 3 days) after the last dose of study drug, Safety Follow up: 90-day (±7 days) after the end-of treatment visit)
  Incidence of anti-drug antibody (ADA) (including serum titers of anti-IMC-001 antibodies) The percentage of patients demonstrating anti-IMC-001 antibodies will be calculated.
Characterize the immunogenicity of IMC-001 : Correlation Between ADA and Drug Exposure and Activity | Screening, prior to infusion at Cycle 4, 7, 10, and 13, End of Treatment, Safety Follow up (each cycle is 14 days, EOT: 28-day (+ 3 days) after the last dose of study drug, Safety Follow up: 90-day (±7 days) after the end-of treatment visit)
  Correlation Between ADA and Drug Exposure and Activity The Spearman nonparametric correlation coefficient will be calculated to quantify the relationship between titer of anti-IMC-001 antibodies and exposure and activity.

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, Principal Investigator — Samsung Medical Center, Republic of Korea
Locations (5):
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Gwangju
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No